CLINICAL TRIAL: NCT04385485
Title: Passive Mobilization With Place and Hold Versus Active Motion Therapy After Flexor Tendon Repair: 5-year Minimum Follow-up of A Randomized Controlled Trial
Brief Title: Passive Mobilization With Place and Hold vs Active Mobilization Therapy After Flexor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Sara Chevalley, Specialist in Hand Surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2017-07-04; First posted 2020-05-13 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Tendon Injury - Hand
Keywords: Flexor tendon injury; Early Mobilisation

STUDY DESIGN:
Intervention Model Description: The Patients are randomised 1-3 days after surgery to either active or passive mobilisation. The randomisation was done by a statistical software program (Medstat) and the protocols are placed in numbered sealed envelopes.
Who Masked: Outcomes Assessor
Masking Description: The occupational therapist who do the evaluation and make all the measurements 6 and 12 months after surgery don't know if the patient was randomised to active or passive mobilisation. Likewise the hand surgeon who do all the measurements at minimum 5 years after surgery don't know which rehabilitation protocol the patient followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active mobilisation (Experimental): The patient see an occupational therapist 1-3 days after surgery. A splint is made to immobilise the wrist and work as a extension block for the MCP-joints. This splint has to be worn day and night for 4 weeks. Another splint that immobilise the distal interphalangeal (DIP) joint and the proximal interphalangeal (PIP) joints are worn whenever the patient is not exercising. During active exercise the patient follows a strict protocol with both active and passive training and increasing number of repetitions. The rehabilitation is proceeding for 3 months.
  Interventions: Procedure: Active mobilisation
- Passive mobilisation with place and hold (Active Comparator): 1-3 days after surgery the patient gets a new plaster that immobilise the wrist and work as an extension block for the MCP-joints. The occupational therapist attach rubberbands to the nails of all the fingers and the training is done passively with active hold according to a strict protocol. The training with rubberbands is done during 4 weeks. After that the rehabilitation is active. The rehabilitation is proceeding for 3 months.
  Interventions: Procedure: Passive mobilisation with place and hold

INTERVENTIONS:
Procedure: Active mobilisation — We investigate if active mobilisation is as good as passive mobilisation with place and hold after flexor tendon suture.
  Arms: Active mobilisation
Procedure: Passive mobilisation with place and hold — We investigate if active mobilisation is as good as passive mobilisation with place and hold after flexor tendon suture.
  Arms: Passive mobilisation with place and hold

SUMMARY:
The aim of this study is to investigate if active mobilisation after flexor tendon repair in fingers gives better range of motion, strength, risk of rupture and patient satisfaction compared with passive mobilisation with place and hold after flexor tenon repair.

DETAILED DESCRIPTION:
Patients with an injury in flexor digitorum profundus (FDP) are eligible for inclusion in this study. The patients are referred to the Department of Hand Surgery at Sahlgrenska University Hospital. Potential patients are informed about the study. An informed consent is obtained from those who accept to participate. The surgery is performed in the same way for all patients with a four-stranded core suture and an epitendinous suture. The randomisation is performed after surgery when the patient is starting up rehabilitation 1-3 days after surgery. The randomisation was done by a computer program and the two different mobilisation protocols are placed accordingly in sealed envelopes numbered from 1 to 64. The envelopes are used one after another in a consecutive order.

All the operations are done by specialists in hand surgery or experienced residents in hand surgery at the clinic. The FDP tendon is repaired with a four-stranded core suture with a 4-0 Ti-cron (nonabsorbable braided polyester) and a running epitendinous suture according to Silfverskiöld with a 6-0 Prolene (nonabsorbable monofil polypropylene). Any concomitant injury in the flexor digitorum superficialis (FDS) tendon is repaired according to the surgeons preference. Any digital nerve is repaired with microsurgical instruments and a 8-0 or 9-0 S&T (non-absorbable polyamide monofilament).

Mobilisation

1-3 days after surgery the patient will be randomised to either active mobilisation or passive mobilisation with rubber bands and active place-and-hold at the hand rehabilitation unit in our clinic. The patients in both groups are closely followed by an occupational therapist for 12 weeks. Additional follow-up appointments are planned after 6 and 12 months. Patients in both groups are allowed to do all kinds of normal activity after 3 months and heavy manual work and gym training after 4 months.

Active mobilisation The active mobilisation program is based on the two programs, Belfast (ref) and Billericay (ref). Our program is a mix between these two. On the first day of mobilisation (1-3 days after surgery) the dressings are changed and a dorsal splint with the wrist in neutral position and the metacarpophalangeal (MCP) joints in 60-80 degrees of flexion is made for the patient. Another removable volar plate keeping the fingers extended is used in addition to the dorsal splint between training sessions.

The patient is instructed to flex the fingers passively with the other hand and then keep the fingers in flexion and do the place and hold for 3 seconds. Then the fingers are extended actively as far as the splint allows. This motion is done with 5 repetitions, 10 times per day with 1.5 hour resting period between sessions. Every second training session (i.e. every third hour) all fingers are flexed actively three times. After a week both the passive motion with place-and-hold and the true active motion is done with 10 repetitions, 10 times per day with a resting time of 1.5 hours between training sessions. Four weeks post surgery flexion and extension of the wrist is added with 10 repetitions, 4 times per day and joint-by-joint training for the injured finger with 3 repetitions 10 times per day in addition to the previous protocol.

Passive mobilisation with place-and-hold Before the mobilisation starts the patients get their dressings changed and a new dorsal forearm plaster ending at the level of the proximal interphalangeal (PIP) joints with the wrist in neutral position and a dorsal block over the proximal phalanges creating an extension block for the MCP-joints of 60-80 degrees. Rubberbands are attached to all the fingernails and a small hook is fastened to the plaster to hang the rubberbands on creating a resting position for the fingers between training sessions. A night splint with the interphalangeal joints in extension is also made to protect the fingers and keep them in full extension when the patient sleeps.

The patient is instructed to flex the fingers passively with the other hand one at a time and then keep the fingers in flexion and do a gentle squeeze, so called place-and-hold. Then the fingers are extended actively as far as the plaster allows. For four weeks the patient do this exercise with 10 repetitions, 10 times a day (7-8 repetitions on the first day) with a resting period of 1.5 hours between sessions. After four weeks the plaster is removed and replaced by a splint protecting the wrist in neutral position and the patient adds true active flexion of the fingers to the previous program with 10 repetitions 10 times per day. Six weeks post surgery the splint is removed and flexion and extension of the wrist is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Primary, complete injury to FDP in digit II-V
* Injury in zone I och II
* Operation within 72 hours from injury
* The patient must be able to fulfill the rehabilitation program.

Exclusion Criteria:

* Concomitant fracture
* Concomitant soft tissue defect
* Severe crush injury
* Palmar plate injury demanding immobilisation
* Concomitant joint injury
* Concomitant extensor tendon injury
* Bilateral injury
* Previous loss of function in the finger before the injury
* Uncertainty if the patient can fulfill the rehabilitation
* The surgeon think it is unsuitable with active training after surgery

Concomitant injury of the flexor digitorum superficialis (FDS) or a digital nerve is accepted. A distal injury in zone I is not included if it requires a reinsertion of the tendon to the bone.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Range of motion | Up to minimum 5 years after surgery
  Range of motion in the proximal and distal interphalangeal joints in the injured finger and corresponding finger in the other hand are measured after 4, 8 and 12 weeks and after 6 and 12 months and minimum 5 years after surgery. We are interested to learn if there is a difference in range of motion between the two study groups.

SECONDARY OUTCOMES:
Jamar grip strength | Up to minimum 5 years after surgery
  Grip strength is measured with a Jamar hydraulic hand dynamometer at 6 and 12 months and minimum 5 years after surgery. We are interested to learn if there is a difference in range of motion between the two study groups.
Key Pinch strength | Up to minimum 5 years after surgery
  Key pinch strength is measured with a hydraulic pinch gauge dynamometer at 6 and 12 months and minimum 5 years after surgery. We are interested to learn if there is a difference in range of motion between the two study groups.
Tendon rerupture | Up to minimum 5 years after surgery
  We record any reruptures continuously during the study period. If there are 3 consecutive reruptures in the active group the study is terminated immediately.
Need of secondary operation | Up to minimum 5 years after surgery
  At 6 and 12 months and minimum 5 years the need for secondary surgery is evaluated
Disabilities of the Arm, Shoulder and Hand (DASH) outcome measure questionaire | Up to minimum 5 years after surgery
  DASH is an outcome questionnaire with 30 questions about functions and symptoms in the upper extremity, answered by the patient. Scores range from 0 (no disability) to 100 (completely disabled). The patients are given the DASH questionaries to fill in before surgery as a baseline and again after 3, 6 and 12 months and minimum 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fridén, Professor, Study Director — Sahlgrenska University Hospital
Locations (1):
- Department of Hand Surgery, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No